CLINICAL TRIAL: NCT01051401
Title: Statin Therapy as a Protective Technique for Potential Cardiovascular Event Occurrences Among Breast Cancer Patients Undergoing Chemotherapy Treatment
Brief Title: Rosuvastatin in Treating Women With Cardiovascular Complications Who Are Undergoing Chemotherapy For Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00009933; NCI-2010-00125 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 98509 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Cardiovascular Complications; Recurrent Breast Cancer; Stage I Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (rosuvastatin) (Experimental): Patients receive rosuvastatin PO once daily for 3 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: rosuvastatin; Other: survey administration; Procedure: management of therapy complications
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO once daily for 3 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: placebo; Other: survey administration; Procedure: management of therapy complications

INTERVENTIONS:
Drug: rosuvastatin — Given PO
  Arms: Arm I (rosuvastatin)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: survey administration — Correlative study
Procedure: management of therapy complications
  Other Names: complications of therapy, management of

SUMMARY:
This randomized pilot clinical trial studies rosuvastatin in treating women with cardiovascular complications who are undergoing chemotherapy for breast cancer. Rosuvastatin may prevent or lessen cardiovascular complications in patients undergoing chemotherapy for breast cancer

DETAILED DESCRIPTION:
OBJECTIVES:

I. Evaluate the feasibility of administering Rosuvastatin to breast cancer patients undergoing treatment with anthracyclines, paclitaxel, cyclophosphamide, and trastuzumab for breast cancer.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive rosuvastatin orally (PO) once daily for 3 months in the absence of disease progression or unacceptable toxicity.

Arm II: Patients receive placebo PO once daily for 3 months in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

Women receiving therapy for breast cancer without a history of cardiovascular disease An low-density lipoprotein (LDL) cholesterol level of less than 160 mg per deciliter (3.4 MMol per liter) Willingness to participate for the duration of the trial (3 months) Written informed consent Triglyceride level of less than 500 mg per deciliter (5.6 mmol per liter)

Exclusion Criteria:

Previous or current use of lipid-lowering therapy Current use of postmenopausal hormone-replacement therapy Evidence of hepatic dysfunction (an alanine aminotransferase level that was more than twice the upper limit of the normal range) Creatine kinase level that was more than three times the upper limit of the normal range Creatinine level that was higher than 2.0 mg per deciliter (176.8 umol per liter) Diabetes Uncontrolled hypertension (systolic blood pressure > 190 mm Hg or diastolic blood pressure > 100 mm Hg) Uncontrolled hypothyroidism (a thyroid-stimulating hormone level that was more than 1.5 times the upper limit of the normal range) Recent history of alcohol or drug abuse or another medical condition that might compromise safety or the successful completion of the study Exclude patients with inflammatory conditions such as severe arthritis, lupus, or inflammatory bowel disease, and patients taking immunosuppressant agents such as cyclosporine, tacrolimus, azathioprine, or long-term oral glucocorticoids Pregnant women are excluded from participation in this study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Whether the rate of statin adherence for patients taking chemotherapy is comparable to the rate of adherence found in prior studies (i.e., JUPITER study) | 3 months

SECONDARY OUTCOMES:
Changes in fasting cholesterol and other patient level characteristics (such as heart rate, blood pressure etc) | At baseline
Changes in fasting cholesterol and other patient level characteristics (such as heart rate, blood pressure etc) | 3 months
Rates of side-effects in the two groups | After 3 months

CONTACTS AND LOCATIONS:
Overall Officials: William Hundley, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States